CLINICAL TRIAL: NCT04638829
Title: Prospective, Multi-center, Open-label Study Measuring Safety and Treatment Satisfaction in Adult Subjects With Chronic Immune Thrombocytopenia (ITP) After Switching to Avatrombopag From Eltrombopag or Romiplostim
Brief Title: Safety and Treatment Satisfaction in Adults With Chronic ITP After Switching to Avatrombopag From Eltrombopag or Romiplostim
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sobi, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AVA-ITP-401
Record Dates: First submitted 2020-11-11; First posted 2020-11-20 (Actual); Results first posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2024-12

CONDITIONS: Immune Thrombocytopenia
Keywords: ITP
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — avatrombopag

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Avatrombopag (Other): Avatrombopag 20 mg oral tablet formulation for 90 days
  Interventions: Drug: Avatrombopag Oral Tablet

INTERVENTIONS:
Drug: Avatrombopag Oral Tablet — Avatrombopag 20 mg given daily for 90 days. Initial dose and dose adjustments will be determined by the physician along with the Doptelet prescribing information
  Other Names: Doptelet

SUMMARY:
Evaluate the safety and tolerability of avatrombopag given for 90 days after stopping treatment with eltrombopag or romiplostim.

DETAILED DESCRIPTION:
This Phase 4, prospective, multi-center, open-label study will evaluate safety, platelet count, and subject reported medication satisfaction in adult subjects with chronic ITP after switching to avatrombopag from eltrombopag or romiplostim. At least 100 subjects will be enrolled, 50 (±10) who have received eltrombopag and 50 (±10) who have received romiplostim for at least 90 days prior to study entry.

ELIGIBILITY:
Inclusion Criteria:

* Subject has been undergoing treatment for primary ITP with eltrombopag or romiplostim for at least 90 days prior to the Screening Visit/Visit 1.
* Subject has had a previous response (at any time) to either eltrombopag or romiplostim, defined as at least 2 platelet counts ≥50×10⁹/L. Subject is willing and able to comply with all aspects of the protocol, including completing the self-administered Treatment Satisfaction Medication Questionnaire (TSQM).

Exclusion Criteria:

* Subject is currently receiving chemotherapy or radiation for any form of cancer.
* Subject with conditions that are likely to prevent them from accurately and reliably completing study assessments, including evidence of moderate to severe dementia, and/or severe and progressive medical illness, as determined by the Investigator.
* Any previous avatrombopag use.
* Previous participation in this study; a subject may not re-enroll after prior discontinuation or completion.
* Enrollment in another clinical study with any investigational drug or device within 30 days of Baseline (or 5 half-lives, whichever is longer); however, participation in observational studies within the previous 30 days is permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2024-01-03 (Actual); Study Completion 2024-01-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (20):
- United States (20):
  - Sobi Site 110, Tucson, Arizona
  - Sobi Site 119, Whittier, California
  - Sobi Site 123, Washington D.C., District of Columbia
  - Sobi Site 129, Miami, Florida
  - Sobi Site 120, Ocala, Florida
  - Sobi Site 125, St. Petersburg, Florida
  - Sobi Site 118, Tampa, Florida
  - Sobi Site 126, Chicago, Illinois
  - Sobi Site 109, Peoria, Illinois
  - Sobi Site 124, New Orleans, Louisiana
  - Sobi Site 101, Bethesda, Maryland
  - Sobi Site 103, Lincoln, Nebraska
  - Sobi Site 121, Chapel Hill, North Carolina
  - Sobi Site 116, Greenville, North Carolina
  - Sobi Site 128, Cleveland, Ohio
  - Sobi Site 127, Philadelphia, Pennsylvania
  - Sobi Site 102, York, Pennsylvania
  - Sobi Site 104, Rock Hill, South Carolina
  - Sobi Site 113, Dallas, Texas
  - Sobi Site 108, Salt Lake City, Utah

REFERENCES:
- [Derived] Tarantino MD, Mosalpuria K, Kolodny S, Zhang J, Vredenburg M, Jamieson BD. Safety, efficacy, and treatment satisfaction in adults with ITP who switched to avatrombopag from another TPO-RA. Blood Adv. 2025 Jun 10;9(11):2733-2743. doi: 10.1182/bloodadvances.2024015635. PMID 40101243

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Avatrombopag
Started | 60
Completed | 57
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Avatrombopag
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.0 (21.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13
  Not Hispanic or Latino | 46
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 5
  White | 43
  More than one race | 1
  Unknown or Not Reported | 8

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability (Adverse Events)
Description: Safety and Tolerability of Avatrombopag given for 90 days after stopping eltrombopag or romiplostim
  The incidence and severity of adverse events (AEs), serious adverse events (SAE) and adverse events of special interest (AESIs) will be summarized for all enrolled subjects using counts and percentages. Treatment-emergent AEs and SAEs will be summarized overall, by system organ class, and by preferred term. AESIs will be summarized by event type (thromboembolic events and bleeding events). In addition, treatment-emergent AEs will be summarized by severity and by relationship to study drug.
  Bleeding events reported during the study will be summarized by WHO grade.
Time Frame: Screening through Day 90 or End of Study
Population: All enrolled subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Avatrombopag
Number analyzed (Participants) | 60
Participants
  TEAEs | 35
  SAEs | 6
  AESIs | 1
  Related TEAEs | 15
  Severe TEAEs | 8
  TEAEs leading to study drug discontinuation | 2

2. Secondary Outcome: Change From Baseline TSQM Convenience Domain Score
Description: Evaluate the change in subject reported outcomes (TSQM - Treatment Satisfaction Questionnaire for Medication) from Baseline. Convenience domain score ranges from 0 to 100, and a higher score indicates a better outcome. Mean Difference was computed as Day 90 minus Baseline and, therefore, a positive mean difference indicates an increase in the score from Baseline to Day 90.
Time Frame: Day 90
Population: All enrolled subjects.
Measure: Mean (95% Confidence Interval); unit: Mean difference in convenience score
Arm/Group | Avatrombopag
Number analyzed (Participants) | 60
Mean difference in convenience score | 13.5 [6.9 to 20.1]
Statistical Analysis 1: Comparison: Avatrombopag; Test type: Other; p = 0.0001, t-test, 2 sided

3. Secondary Outcome: Change From Baseline TSQM Side Effects Domain Score
Description: Evaluate the change in subject reported outcomes (TSQM - Treatment Satisfaction Questionnaire for Medication) from Baseline. Side Effects domain score ranges from 0 to 100, and a higher score indicates a better outcome. Mean Difference was computed as Day 90 minus Baseline and, therefore, a positive mean difference indicates an increase in the score from Baseline to Day 90.
Time Frame: Day 90
Measure: Mean (95% Confidence Interval); unit: Mean difference in side effects score
Arm/Group | Avatrombopag
Number analyzed (Participants) | 60
Mean difference in side effects score | 8.3 [2.1 to 14.4]
Statistical Analysis 1: Comparison: Avatrombopag; Test type: Other; p = 0.0093, t-test, 2 sided

4. Secondary Outcome: Change From Baseline TSQM Effectiveness Domain Score
Description: Evaluate the change in subject reported outcomes (TSQM - Treatment Satisfaction Questionnaire for Medication) from Baseline. Effectiveness domain score ranges from 0 to 100, and a higher score indicates a better outcome. Mean Difference was computed as Day 90 minus Baseline and, therefore, a positive mean difference indicates an increase in the score from Baseline to Day 90.
Time Frame: Day 90
Measure: Mean (95% Confidence Interval); unit: Mean difference in effectiveness score
Arm/Group | Avatrombopag
Number analyzed (Participants) | 60
Mean difference in effectiveness score | 14.4 [7.0 to 21.8]
Statistical Analysis 1: Comparison: Avatrombopag; Test type: Other; p = 0.0003, t-test, 2 sided

5. Secondary Outcome: Change From Baseline TSQM Global Satisfaction Domain Score
Description: Evaluate the change in subject reported outcomes (TSQM - Treatment Satisfaction Questionnaire for Medication) from Baseline. Global Satisfaction domain score ranges from 0 to 100, and a higher score indicates a better outcome. Mean Difference was computed as Day 90 minus Baseline and, therefore, a positive mean difference indicates an increase in the score from Baseline to Day 90.
Time Frame: Day 90
Measure: Mean (95% Confidence Interval); unit: Mean difference in global satisfaction
Arm/Group | Avatrombopag
Number analyzed (Participants) | 60
Mean difference in global satisfaction | 14.2 [8.8 to 19.5]
Statistical Analysis 1: Comparison: Avatrombopag; Test type: Other; p < 0.0001, t-test, 2 sided

6. Secondary Outcome: Proportion of Subjects Who Have a Platelet Count Between ≥50×10^9/L to ≤200×10^9/L
Time Frame: Day 15
Population: All enrolled subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Avatrombopag
Number analyzed (Participants) | 60
Participants | 19

7. Secondary Outcome: Proportion of Subjects Who Have a Platelet Count Between ≥50×10^9/L to ≤200×10^9/L
Time Frame: Day 30
Measure: Count of Participants; unit: Participants
Arm/Group | Avatrombopag
Number analyzed (Participants) | 60
Participants | 33

8. Secondary Outcome: Proportion of Subjects Who Have a Platelet Count Between ≥50×10^9/L to ≤200×10^9/L
Time Frame: Day 60
Measure: Count of Participants; unit: Participants
Arm/Group | Avatrombopag
Number analyzed (Participants) | 60
Participants | 36

9. Secondary Outcome: Proportion of Subjects Who Have a Platelet Count Between ≥50×10^9/L to ≤200×10^9/L
Time Frame: Day 90
Measure: Count of Participants; unit: Participants
Arm/Group | Avatrombopag
Number analyzed (Participants) | 60
Participants | 33

ADVERSE EVENTS:
Time Frame: 90 days
Arm/Group | Avatrombopag
All-Cause Mortality (participants affected / at risk) | 1/60
Serious Adverse Events (participants affected / at risk) | 6/60
Other Adverse Events (participants affected / at risk) | 34/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Avatrombopag (N=60)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2)
Rectal Haemorrhage (Gastrointestinal disorders) | 1 (1)
Sudden Death (General disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Avatrombopag (N=60)
Headache (Nervous system disorders) | 8 (13)
Contusion (Injury, poisoning and procedural complications) | 7 (7)
Oedema Peripheral (General disorders) | 4 (4)
COVID-19 (Infections and infestations) | 3 (3)
Dizziness (Ear and labyrinth disorders) | 3 (3)
Fatigue (General disorders) | 3 (5)
Peripheral Swelling (General disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (3)
Pain (General disorders) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PIs are not allowed to publish clinical trial data on their own after trial completion.

DOCUMENTS (2):
  • Study Protocol (2022-01-28): https://cdn.clinicaltrials.gov/large-docs/29/NCT04638829/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-31): https://cdn.clinicaltrials.gov/large-docs/29/NCT04638829/SAP_001.pdf